CLINICAL TRIAL: NCT07175272
Title: Evaluation of The Effect of Holy Basil in The Treatment of Patients With Dyspepsia
Brief Title: Holy Basil in The Treatment of Dyspepsia
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Watcharasak Chotiyaputta, Associate Professor, Mahidol University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Si 643/2025
Record Dates: First submitted 2025-09-09; First posted 2025-09-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Dyspepsia and Other Specified Disorders of Function of Stomach
Keywords: Dyspepsia; Gastritis; Holy basil
MeSH Terms: conditions — Dyspepsia; Gastritis | interventions — holy basil leaf extract

STUDY DESIGN:
Intervention Model Description: This is a single-center, open-label, single-arm clinical trial designed to evaluate the effects of holy basil extract in adults with dyspepsia. All eligible participants will receive 300 mg of holy basil extract orally once daily for 28 days. Outcomes will be assessed by comparing baseline and post-treatment measures within the same participants.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Holy basil (Experimental): All participants will receive holy basil extract 300 mg orally once daily for 28 days.
  Interventions: Drug: Holy basil extract

INTERVENTIONS:
Drug: Holy basil extract — Holy basil extract (Ocimum sanctum) will be provided as an oral capsule formulation. Each capsule contains 300 mg of standardized holy basil extract with defined amounts of active compounds including ursolic acid (≥0.10 mg) and rosmarinic acid (≥0.50 mg). Participants will be instructed to take one capsule once daily for 28 consecutive days.
  The capsules will be dispensed in blister packs, with labeling according to clinical trial regulatory requirements. Participants will be asked to record daily intake in a study diary, and compliance.

SUMMARY:
The goal of this clinical trial is to evaluate whether holy basil extract can reduce gastric inflammation and improve symptoms in adult patients with dyspepsia.

The main questions it aims to answer are:

* Does holy basil extract reduce gastric mucosal inflammation as measured by histopathology?
* Does holy basil extract improve dyspeptic symptoms, endoscopic findings, gastric pH, duodenal eosinophil counts, and systemic inflammation (serum IL-6)?

Participants will:

* Take 300 mg of holy basil extract orally once daily for 28 days
* Complete symptom questionnaires and diaries during treatment
* Undergo upper endoscopy with biopsy and intragastric pH monitoring before and after treatment
* Provide blood samples for inflammatory marker measurement
* Be monitored for safety and adverse events

DETAILED DESCRIPTION:
Functional dyspepsia is a common condition that causes chronic upper abdominal discomfort, bloating, and early satiety in the absence of structural disease. Conventional therapies such as acid suppression medications or prokinetics provide incomplete symptom relief for many patients, and newer approaches are needed. Increasing evidence suggests that mucosal inflammation, duodenal eosinophilia, and systemic immune activation may play a key role in the disorder.

Holy basil (Ocimum sanctum), or tulsi, is a traditional medicinal herb with anti-inflammatory and gastroprotective properties demonstrated in preclinical studies. It has been shown to reduce gastric acid secretion, increase mucus production, and decrease inflammatory cell infiltration in animal models, but its clinical effects in patients with dyspepsia have not been studied.

This single-center, open-label trial will enroll 27 adults with dyspeptic symptoms at Siriraj Hospital, Mahidol University. All participants will receive 300 mg of holy basil extract once daily for 28 days. The primary outcome is the change in gastric mucosal inflammation assessed by histopathology before and after treatment. Secondary outcomes include improvement in dyspeptic and reflux symptoms, reduction in duodenal eosinophil counts, changes in gastric mucosal appearance on endoscopy, alterations in intragastric pH, and changes in serum interleukin-6 levels as a marker of systemic inflammation. Safety and tolerability will also be evaluated.

Participants will undergo baseline evaluations, including symptom assessment, blood tests, 24-hour pH monitoring, and upper endoscopy with biopsy. These procedures will be repeated at the end of the 28-day treatment period. Weekly monitoring will include review of symptoms, adverse events, and medication compliance.

The study is designed to provide clinical evidence on whether holy basil extract can improve gastric inflammation and relieve symptoms in patients with dyspepsia. Results may support its role as a novel herbal-based therapy for functional dyspepsia.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged 18 years and older.
* Presence of dyspeptic symptoms, assessed by the Leeds Dyspepsia Questionnaire with a score of at least 5 or higher.

Exclusion Criteria:

* Presence of Helicobacter pylori infection.
* Diagnosis of peptic ulcer or erosive esophagitis Los Angeles Classification grade B or greater.
* Use of acid-suppressant therapy including proton pump inhibitors (PPIs) or histamine-2 receptor antagonists (H2RAs) that cannot be discontinued at least 2 weeks prior enrolment and during the study period.
* Use of mucosal protective agents, such as rebamipide, sucralfate, or irsogladine that cannot be discontinued at least 4 weeks prior enrolment and during the study period.
* History of gastric cancer or duodenal cancer.
* Previous upper gastrointestinal surgery.
* Current pregnancy or lactation.
* Known allergic to the medicine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in gastric mucosal inflammation score by histopathology | From baseline to the end of treatment at 28 days
  Degree of gastric mucosal inflammation assessed by histopathological examination using the Updated Sydney System, measured at baseline and after 28 days of treatment.

SECONDARY OUTCOMES:
Change in dyspeptic symptoms | From baseline to the end of treatment at 28 days
  Dyspeptic symptoms such as epigastric pain, fullness, bloating, and nausea will be assessed using the Leeds Dyspepsia Questionnaire. Total and individual symptom scores will be recorded at baseline and after 28 days of treatment, and changes will be analyzed.
Change in gastroesophageal reflux symptoms | From baseline to the end of treatment at 28 days
  Symptoms of gastroesophageal reflux disease, including heartburn and regurgitation, will be evaluated using the Frequency Scale for the Symptoms of GERD (FSSG). Scores will be compared between baseline and post-treatment assessments.
Change in gastric mucosal appearance | From baseline to end of treatment at 28 days
  Endoscopic appearance of the gastric mucosa will be assessed using the Modified Lanza Score (MLS) during upper endoscopy. The severity of gastric mucosal injury will be graded, and scores will be compared before and after treatment.
Change in duodenal eosinophil count | From baseline to end of treatment at 28 days
  Biopsies from the duodenum will be examined histologically to determine intraepithelial eosinophil counts. The mean number of eosinophils per high-power field will be compared between baseline and after 28 days of holy basil extract.
Change in intragastric pH | From baseline to end of treatment at 28 days
  Gastric acid levels will be assessed by 24-hour ambulatory intragastric pH monitoring. Mean pH values and time spent below pH thresholds will be recorded and compared between baseline and after treatment.
Change in esophageal acid exposure time | From baseline to end of treatment at 28 days
  Esophageal acid exposure will be assessed by 24-hour ambulatory pH monitoring. Mean pH values and time spent below pH thresholds will be recorded and compared between baseline and after treatment.
Change in serum interleukin-6 (IL-6) levels | From baseline to end of treatment at 28 days
  Blood samples will be collected to measure serum IL-6 levels as a marker of systemic inflammation. Baseline values will be compared to those after 28 days of treatment.
Incidence of adverse events | From baseline to end of treatment at 28 days
  All adverse events and side effects reported by participants or observed by investigators will be collected, categorized by severity and relationship to study medication, and summarized.

CONTACTS AND LOCATIONS:
Overall Officials: Monthira Maneerattanaporn, MD, Principal Investigator — Mahidol University; Somchai Leelakusolvong, MD, Study Chair — Mahidol University; Tanawat Geeratragool, MD, Study Chair — Mahidol University; Pubet Weeranawin, MD, Study Chair — Mahidol University
Locations (1):
- Faculty of Medicine Siriraj Hospital, Mahidol University, Bangkok Noi, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No
To protect participant confidentiality and comply with institutional and regulatory requirements, no IPD will be shared unless with reasonable request.

REFERENCES:
- [Background] Jamshidi N, Cohen MM. The Clinical Efficacy and Safety of Tulsi in Humans: A Systematic Review of the Literature. Evid Based Complement Alternat Med. 2017;2017:9217567. doi: 10.1155/2017/9217567. Epub 2017 Mar 16. PMID 28400848
- [Background] Dharmani P, Kuchibhotla VK, Maurya R, Srivastava S, Sharma S, Palit G. Evaluation of anti-ulcerogenic and ulcer-healing properties of Ocimum sanctum Linn. J Ethnopharmacol. 2004 Aug;93(2-3):197-206. doi: 10.1016/j.jep.2004.02.029. PMID 15234753
- [Background] Pattanayak P, Behera P, Das D, Panda SK. Ocimum sanctum Linn. A reservoir plant for therapeutic applications: An overview. Pharmacogn Rev. 2010 Jan;4(7):95-105. doi: 10.4103/0973-7847.65323. PMID 22228948
- [Background] Wauters L, Talley NJ, Walker MM, Tack J, Vanuytsel T. Novel concepts in the pathophysiology and treatment of functional dyspepsia. Gut. 2020 Mar;69(3):591-600. doi: 10.1136/gutjnl-2019-318536. Epub 2019 Nov 29. PMID 31784469
- [Background] Ford AC, Moayyedi P, Black CJ, Yuan Y, Veettil SK, Mahadeva S, Kengkla K, Chaiyakunapruk N, Lee YY. Systematic review and network meta-analysis: efficacy of drugs for functional dyspepsia. Aliment Pharmacol Ther. 2021 Jan;53(1):8-21. doi: 10.1111/apt.16072. Epub 2020 Sep 16. PMID 32936964